CLINICAL TRIAL: NCT03149458
Title: Effects of a Dance Workshop on the Balance Abilities of Hemiparetic Patients
Brief Title: Dance Workshop on Balance of Hemiparetic Patients
Acronym: DanceStudio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Fondation Garches (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01876-45
Record Dates: First submitted 2017-02-27; First posted 2017-05-11 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Hemiparesis
Keywords: stroke; balance; dance
MeSH Terms: conditions — Paresis; Stroke

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance group (Experimental): dance program for 8 one-hour sessions.
  Interventions: Other: dance
- control group (Active Comparator): upper limb rehabilitation for 8 one-hour sessions.
  Interventions: Other: control

INTERVENTIONS:
Other: dance — dance program
  Arms: Dance group
Other: control — upper limb rehabilitation
  Arms: control group

SUMMARY:
The majority of hemiparetic patients have balance disorders, which impact independence in daily living activities and walking. Conventional techniques used in rehabilitation improve balance but have shown no effects on dynamic balance required during walking. Recently dance is proposed to improve dynamic balance in older people and people with Parkinson's disease. Although many studies showed that dance is an effective activity to improve balance in these people, it has never been assessed in hemiparetic patients (except a case report). The aim of this study is to show that a dance program improves the balance of hemiparetic patients, compared to a control group. This randomized controlled study aims to include 40 hemiparetic patients who will perform a dance program (experimental group) or a upper-limb rehabilitation program (control group) for 8 one-hour sessions.

DETAILED DESCRIPTION:
Randomized controlled study aims to include 40 hemiparetic patients who will perform a dance program (experimental group) or a upper-limb rehabilitation program (control group) for 8 one-hour sessions. These activities are carried out in the form of a workshop and are already proposed in common practice in the service. They are carried out by the physiotherapists of the service. Patients are assigned in one of two study groups. It is specified that they will be able to carry out the program of the opposing group at the end of the study in order to limit the "disappointment" effect. The evaluations will be carried out at 4 and 8 weeks and will mainly rely on data of balance, function, quality of life and satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Patient who signed the consent letter
* Male or female adults age ≥ 18 years,
* Hemiparetic patient
* Patient with balance disorders, able to walk alone and perform a U-turn, with or without technical assistance.

Exclusion Criteria:

* Bilateral brain lesions, cerebellar syndrome
* Other pathology or impairment that may interfere with the study such as visual, cardiovascular or other uncontrolled medical conditions
* Patient who underwent surgery of the musculoskeletal system in The 6 months prior to inclusion
* Major cognitive disorders not allowing the dance activity or the passing of evaluations
* Behavioral disorders not allowing group workshops
* Pregnant woman, breastfeeding
* Non-affiliation to a social security scheme (beneficiary or beneficiary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Timed up and Go | 5min
  get up, walk 3m, turn around and return sit down

SECONDARY OUTCOMES:
Berg Balance Scale | 10min
  clinical scale assessing balance. 14-item scale designed to measure balance of the older adult in a clinical setting. Scoring: A five-point scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Total Score = 56

CONTACTS AND LOCATIONS:
Overall Officials: François GENET, PhD, Principal Investigator — Centre d'Investigation Clinique et Technologique 805
Locations (1):
- Raymond Poincaré Hospital- PMR Unit - Netter, Garches, France

IPD SHARING:
Plan to Share IPD: No